CLINICAL TRIAL: NCT06134089
Title: Evaluating Online Messages About Colon Cancer Screening
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: HCI164736
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Colonic Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perceived Shareablility Prompt First
  Interventions: Behavioral: Perceived Effectiveness Prompt; Behavioral: Perceived Shareability Prompt
- Perceived Effectiveness Prompt First
  Interventions: Behavioral: Perceived Effectiveness Prompt; Behavioral: Perceived Shareability Prompt

INTERVENTIONS:
Behavioral: Perceived Effectiveness Prompt — Participants will assess pairs of messages with the prompt, "Which of the messages below is more likely to make you want to get screened for colorectal cancer?
  Participants will also be able to provide their own idea for a message rather than selecting a message from the pairs presented.
Behavioral: Perceived Shareability Prompt — Participants will assess pairs of messages with the prompt, "Which of the messages below would you be more likely to share with your friends or family?"
  Participants will also be able to provide their own idea for a message rather than selecting a message from the pairs presented.

SUMMARY:
The goal of the study is to determine, using a choice-based approach, what messages (pulled from various online sites) people find more and less persuasive and shareable on the topic of colorectal cancer screening. As a secondary goal, the study is interested how various information behaviors, such as people's self-reported seeking of health information and encountering of health information, demographic variables, individual difference variables, and message exposure associate with their intentions to adhere to recommended colorectal cancer screening guidelines from the National Cancer Institute. The study is interested at differences specifically among Black and White Americans of recommended screening age (45-74).

ELIGIBILITY:
Inclusion Criteria:

* Identify as white/Caucasian or Black/African American.

Exclusion Criteria:

* Do not identify as white/Caucasian or Black/African American.
* Previously diagnosed with colorectal cancer

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be White (n=1,000) and Black (n=1,000) Americans between the ages of 45 and 74. The goal of the study is to determine if there are differences in message preferences and evaluations between these two groups due to historical disparities in colorectal cancer screening uptake and outcomes.
Sampling Method: Probability Sample
Enrollment: 2210 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy J. King, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- University of Utah Hospital/ Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2210 participants started the study, and 24 participants were removed from the analyzed data.
Groups:
- Perceived Shareablility Prompt First; Perceived Effectiveness Prompt First: Perceived Effectiveness Prompt: Participants will assess pairs of messages with the prompt, "Which of the messages below is more likely to make you want to get screened for colorectal cancer?
  Participants will also be able to provide their own idea for a message rather than selecting a message from the pairs presented.
  Perceived Shareability Prompt: Participants will assess pairs of messages with the prompt, "Which of the messages below would you be more likely to share with your friends or family?"
  Participants will also be able to provide their own idea for a message rather than selecting a message from the pairs presented.
- Undetermined First Message Prompt: These participants were not included in the analysis, as it was not clear if they saw the effectiveness/shareability prompt first.
  As their group assignment could not be determined, the data from these participants were not included in the analysis, as their associated data was deemed unreliable.
Period: Overall Study
Arm/Group | Perceived Shareablility Prompt First | Perceived Effectiveness Prompt First | Undetermined First Message Prompt
Started | 1051 | 1135 | 24
Completed | 1051 | 1135 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the "Undetermined First Message Prompt" group were excluded from baseline characteristics reporting because baseline characteristics data were not available. Data for this group were not collected during the study, as evidenced by blank fields or entries containing erroneous or unusable information. These participants could not be included in the reported dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Perceived Shareablility Prompt First | Perceived Effectiveness Prompt First | Undetermined First Message Prompt | Total
Number analyzed (Participants) | 1051 | 1135 | 0 | 2186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 740 | 783 |  | 1523
  >=65 years | 311 | 352 |  | 663
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.45 (8.12) | 59.52 (8.14) |  | 59.48 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 565 | 640 |  | 1205
  Male | 486 | 495 |  | 981
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 1051 | 1135 |  | 2186
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 525 | 547 |  | 1072
  White | 526 | 588 |  | 1114
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1051 | 1135 |  | 2186

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Determining Messages
Description: This outcome measure will report the number of participants who participated in determining the Online Messages About Colon Cancer Screening. This study will help determine the content of Colon Cancer Screening messaging for future research.
Time Frame: 15 minutes
Population: Participants in the "Undetermined First Message Prompt" group were excluded from outcome measure reporting because data were not available. Data for this group were not collected during the study, as evidenced by blank fields or entries containing erroneous or unusable information. These participants could not be included in the reported dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Perceived Shareablility Prompt First | Perceived Effectiveness Prompt First | Undetermined First Message Prompt
Number analyzed (Participants) | 1051 | 1135 | 0
Participants | 1051 | 1135 | 0

2. Secondary Outcome: Intentions to Follow Screening Recommendations in the Future
Description: Single item self-report of intentions to follow USPSTF recommendations for colorectal cancer screening on a seven-point scale. A low score (Minimum: 1 Extremely Unlikely to follow USPSTF recommendations) is an unfavorable outcome and a high score (Maximum: 7 Extremely Likely to follow USPSTF recommendations) is a favorable outcome.
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Perceived Shareablility Prompt First | Perceived Effectiveness Prompt First | Undetermined First Message Prompt
Number analyzed (Participants) | 1036 | 1127 | 0
units on a scale | 5.65058 (1.94) | 5.65395 (1.935) |

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected for this study.
Description: All-Cause Mortality data was not collected for this study..
Arm/Group | Perceived Shareablility Prompt First | Perceived Effectiveness Prompt First | Undetermined First Message Prompt
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT06134089/Prot_SAP_000.pdf